CLINICAL TRIAL: NCT04652323
Title: Subcutaneous Connective Tissue Reactions to New Calcium Silicate Cements: An Animal Study
Brief Title: Tissue Reactions to Calcium Silicate
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Seçil Çalışkan, Assistant Professor, Eskisehir Osmangazi University
Other Study IDs: 13.02.2019 / 2019-02/04
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Dental Materials; Mineral Trioxide Aggregate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (4):
- Control: Twenty-one empty polyethylene tubes remained empty to bewere used as in the control group.
  Interventions: Drug: Biocompatibility of calcium silicate cements
- ProRoot MTA: ProRoot White MTA mixed according to the manufacturer's' instructions were filled placed into sterile p olyethylene tubules (internal diameter: 1.3 mm internal diameter, x external diameter: 1.6 mm external diameter, x length: 5.0 mm length) sterilized with ethylene oxide gas, as specified by ISO , with using a sterile Llentulo.
  Interventions: Drug: Biocompatibility of calcium silicate cements
- Medcem MTA: Medcem MTA mixed according to the manufacturer's' instructions were filled placed into sterile p olyethylene tubules (internal diameter: 1.3 mm internal diameter, x external diameter: 1.6 mm external diameter, x length: 5.0 mm length) sterilized with ethylene oxide gas, as specified by ISO , with using a sterile Llentulo.
  Interventions: Drug: Biocompatibility of calcium silicate cements
- Medcem Pure Portland Cement: Medcem Pure Portland Cement mixed according to the manufacturer's' instructions were filled placed into sterile p olyethylene tubules (internal diameter: 1.3 mm internal diameter, x external diameter: 1.6 mm external diameter, x length: 5.0 mm length) sterilized with ethylene oxide gas, as specified by ISO , with using a sterile Llentulo.
  Interventions: Drug: Biocompatibility of calcium silicate cements

INTERVENTIONS:
Drug: Biocompatibility of calcium silicate cements — The presence of inflammation, edema, necrosis, dystrophic calcification, and thickness of fibrous capsule formation was recorded by histological examination 7, 30, and 60 days after the implantation procedure of materials.

SUMMARY:
The aim of this study was to determine the subcutaneous connective tissue reactions to these new materials.

Materials and Methods These materials were placed in polyethylene tubes and implanted into the dorsal connective tissue of Sprague Dawley rats. The presence of inflammation, edema, necrosis, dystrophic calcification, and thickness of fibrous capsule formation was recorded by histological examination 7, 30, and 60 days after the implantation procedure. Inflammation scores were defined as follows: 0 = no or few inflammatory cells, no reaction, 1 = <25 cells, mild reaction; 2 = 25 to 125 cells, moderate reaction; and 3 = ≥125 cells, severe reaction. Fibrous capsule thickness, necrosis, and formation of calcification were recorded.

DETAILED DESCRIPTION:
24 Twenty-four male Sprague Dawley rats weighing 250--300 gr were used in the study. For preliminary study, 1 one rat was used on each experimental day . During the study period, the animals were kept in cages in groups of five and taken to daily care under standard care conditions without restriction ofno feed and water supply restrictions.

ProRoot White MTA, Medcem Pure Portland Cement, and Medcem MTA mixed according to the manufacturer's' instructions were filled placed into sterile p olyethylene tubules (internal diameter: 1.3 mm internal diameter, x external diameter: 1.6 mm external diameter, x length: 5.0 mm length) sterilized with ethylene oxide gas, as specified by ISO , with using a sterile Llentulo. Twenty-one empty polyethylene tubes remained empty to bewere used as in the control group.

Surgical Procedures The rats were anesthetized in an ether jar, followed byand then received intraperitoneal administration of 70- mg/kg ketamine and 10- mg/kg xylazine intraperitoneally. The operation area (backs) of the anesthetizedeach rats were was shaved with a certain razor blade, and the surgical area was disinfected with Betadine skin disinfectant ,. After shaving, the operation area wasand covered with sterile drapes to be exposed. In orderTo induce local hemostasis, operations of 0.5 cc, 0.006- mg/ml 4% articaine containing epinephrine (Ultracaine D-S-Aventis Forte, Istanbul, Turkey) by infiltrating local anesthesia was performedadministered.

Incision lines were determined marked on the dorsal, anterior, and posterior extremities of the experimental animals, two in the anterior and two in the posterior region and two in the posterior region. When determining the incision lines, cCare was taken to keep a distance of at least 2 cm distance between the placed materials to prevent them from being affected . Skin iIncisions of approximately 1 cm length long was performedwere made with the a sterile scalpel in the designated areas. The cCanals were entered through the incision site with a sterile periosteal elevator, and ducts were opened under the skin by blunt dissection approximately 2 cm deep. Subsequently, polyethylene tubules filled with the experimental material according toof the each groups and sterile empty polyethylene tubules for the control groups were placed in the prepared subcutaneous canals. The incision sites were then closed primarily using 3/0 silk sutures. Antibacterial spray was applied on the sutures.

Histological Procedures After surgery, on the 7th, 30th and 60th days, 7seven animals from each group, (21 animals) were euthanized intraperitoneally with high doses of thiopentalsodium (Pental, İ.E. Ulagay Med. San. , Istanbul, Turkey) administered intraperitoneally under ether anesthesia on Days 7, 30, and 60. Then, tThe test tubules placed were then removed together with the surrounding tissues and placed in bottles containing 10% neutral formalin. Paraffin blocks were prepared from test samples fixed in bottles containing 10% formalin for 2 two days. From the tissues embedded in the paraffin blocks, 4- μm serial sections parallel to the long axis of the tube were taken cut with a microtome (Leica SM 2000R, Leica Instruments, Wetzlar, Germany) and stained with hematoxylin and eosin (H&E).

All histological evaluations were performed The tissue samples were histologically examined under an optical microscope (Nikon Eclipse E 600, Nikon Corp., Tokyo, Japan) at 40×x, 100×x, 200×x, and 400×x magnifications. All the slides were examined and rated by a pathologists blinded to all procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male Sprague Dawley rats weighing 250--300 gr

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult
Study Population: 24 Twenty-four male Sprague Dawley rats weighing 250--300 gr were used in the study.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Biocompatiblity | 1 year
  determine the subcutaneous connective tissue reactions to ProRoot MTA, Medcem MTA and Medcem Pure Portland Cement

CONTACTS AND LOCATIONS:
Overall Officials: Seçil Çalışkan, Principal Investigator — Eskişehir Osmangazi University
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided